CLINICAL TRIAL: NCT00000352
Title: Effects of Dextromethorphan on Opioid Tolerance in Methadone Patients
Brief Title: Effects of Dextromethorphan on Opioid Tolerance in Methadone Patients - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-1; Y01-3-0012-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1997-08

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan

SUMMARY:
The purpose of this study is to determine if addition of dextromethorphan to a stable dose of methadone in opioid dependent subjects will significantly affect physical and psychological aspects of opioid tolerance.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-12; Primary Completion 1998-02 (Actual); Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States